CLINICAL TRIAL: NCT00769951
Title: The Geriatric-Oncology Database: A Resource for Advancing Research in Older Cancer Patients
Brief Title: Study of Physical and Mental Health of Older Patients With Newly Diagnosed Cancer
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE9Y07
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Cognitive/Functional Effects; Depression; Hematopoietic/Lymphoid Cancer; Malnutrition; Pain; Psychosocial Effects of Cancer and Its Treatment; Unspecified Adult Solid Tumor, Protocol Specific; Weight Changes
Keywords: pain; depression; weight changes; cognitive/functional effects; malnutrition; psychosocial effects of cancer and its treatment; unspecified adult solid tumor, protocol specific; hematopoietic/lymphoid cancer
MeSH Terms: conditions — Depression; Hematologic Neoplasms; Malnutrition; Pain; Body Weight Changes | interventions — Mental Status and Dementia Tests; Psychiatric Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: medical chart review — Data will be obtained from patients medical records at baseline, 6 months, 1 year, and 3 years.
Other: questionnaire administration — Patients undergo a 1-hour comprehensive geriatric assessment at baseline and periodically during the study as part of routine care. The assessments include the Lawton's nine-item Instrumental Activities of Daily Living (IADL); the Katz's Activity of Daily Living (ADL); the Timed Up and Go Test; the Karnofsky Physician-Rated Performance Rating Scale (KPS); the number of falls in the past 6 months; the Mini Nutritional Assessment (MNA); the Body Mass Index; the percent of unintentional weight loss in the past 6 months; the Medical Outcomes Study (MOS) Social Support Subscale (emotional/information and tangible subscales); the MOS Social Activity Limitations Measures; the Charlson Comorbidity Index; the Cumulative Index Rating Scale Geriatrics (CIRS-G); the ACE-27; the Folstein's Mini-Mental State Examination (MMSE); the Geriatric Depression Scale (GDS); the Functional Pain Scale; and a list of medications.
Procedure: cognitive assessment — Patients undergo a 1-hour comprehensive geriatric assessment at baseline and periodically during the study as part of routine care.
Procedure: psychosocial assessment and care — Patients undergo a 1-hour comprehensive geriatric assessment at baseline and periodically during the study as part of routine care.
Procedure: quality-of-life assessment — Patients undergo a 1-hour comprehensive geriatric assessment at baseline and periodically during the study as part of routine care.

SUMMARY:
RATIONALE: Gathering information from older patients with newly diagnosed cancer may help doctors learn more about the risks of functional decline.

PURPOSE: This studying is looking at the physical and mental health of older patients with newly diagnosed cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To create a Geriatric-Oncology database of patients 65 years of age and older with newly diagnosed cancer who have been identified as being at increased risk of functional decline and mortality within a year.
* To enhance the Geriatric-Oncology Database by linking it to the Central Medicare Services (CMS) Database and the Ohio Death Files.

OUTLINE: This is a multicenter study.

Patients undergo a 1-hour comprehensive geriatric assessment at baseline and periodically during the study as part of routine care. The assessments include the Lawton's nine-item Instrumental Activities of Daily Living (IADL); the Katz's Activity of Daily Living (ADL); the Timed Up and Go Test; the Karnofsky Physician-Rated Performance Rating Scale (KPS); the number of falls in the past 6 months; the Mini Nutritional Assessment (MNA); the Body Mass Index; the percent of unintentional weight loss in the past 6 months; the Medical Outcomes Study (MOS) Social Support Subscale (emotional/information and tangible subscales); the MOS Social Activity Limitations Measures; the Charlson Comorbidity Index; the Cumulative Index Rating Scale Geriatrics (CIRS-G); the ACE-27; the Folstein's Mini-Mental State Examination (MMSE); the Geriatric Depression Scale (GDS); the Functional Pain Scale; and a list of medications.

Data will be obtained from patients medical records at baseline, 6 months, 1 year, and 3 years. At completion of 1 and 3 years of follow up, the Geriatric-Oncology Database will be linked to the Central Medicare and Medicaid Services (CMS) Database and the Ohio Death Files.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed cancer

  * Any stage disease
* At increased risk for functional decline and mortality within the next year as per the Vulnerable Elders Survey (VES-13) screening tool (score ≥ 3)
* Seeking care at the Ireland Cancer Center (University hospitals and all other satellite sites)
* Patients with a pre-existing cancer diagnosis and a geriatric syndrome referred directly to the Senior Adult Oncology Program by their providers for a geriatric-oncology consultative evaluation are not eligible

PATIENT CHARACTERISTICS:

* Able to speak and comprehend English
* Able to understand and willing to sign a written informed consent

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Primary care clinics
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2008-02; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Creation of a Geriatric-Oncology database | Data will be obtained from patients medical records at baseline, 6 months, 1 year, and 3 years.
Enhancement of the Geriatric-Oncology database by linking it to the Central Medicare Services Database and the Ohio Death Files | At completion of 1 and 3 years of follow up, the Geriatric-Oncology Database will be linked to the Central Medicare and Medicaid Services (CMS) Database and the Ohio Death Files.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Owusu, MD, MSC, Study Chair — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - UHHS Chagrin Highlands Medical Center, Cleveland, Ohio